CLINICAL TRIAL: NCT02675686
Title: Amniotic Fluid Biomarker Research for Prediction of Postnatal Renal Function in Fetus With a Bilateral Abnormal Renal Development: National, Multicenter, Prospective and Non-interventional Study.
Brief Title: Amniotic Biomarkers for the Prediction of Postpartum Renal Function.
Acronym: BIOMAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 10 138 01; 2010-A01151-38 (Registry Identifier: Agence National du Médicament et des Produits de santé)
Record Dates: First submitted 2015-07-10; First posted 2016-02-05 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Amniotic fluid, obtained during routine clinical management. Whole blood from live born children for renal function determination obtained during routine clinical management.
Oversight: Data Monitoring Committee: No

SUMMARY:
The discovery of antenatal bilateral renal anomaly poses an essential question: can we predict postnatal renal function? Ultrasound is insufficiently precise to predict postnatal renal function evolution.

The objective of this study is to estimate the specificity and sensitivity of amniotic fluid biomarkers to predict postnatal renal function in fetuses with bilateral developmental nephropathies.

Both fetuses with bilateral renal anomalies and control (healthy) fetuses will be included.

For this study amniotic fluid will only be collected according to routine clinical practice and only excess amniotic fluid sample will be used for the study.

The potentially identified biomarkers will not change routine management of the pregnancies in the study.

ELIGIBILITY:
INCLUSION CRITERIA:

All fetuses with a bilateral abnormal renal development (structure modification of the parenchyma with or without urinary tract abnormalities associated)

The following sonographic criteria are used:

* Fetal kidney size <2.5ep or <2 standard deviation (SD) defining renal hypoplasia or renal size> 97.5ep or> 2 SD defining nephromegaly
* And / or hyperechogenicity (more echogenic than the liver kidney)
* And / or cysts
* And / or abnormal cortico-medullary differentiation (decrease or lack thereof)
* And / or bilateral cortical thinning
* And / or the possibility of an initial unilateral renal disease in the case of a pathology on which kidney damage is usually to become bilateral during evolution

EXCLUSION CRITERIA:

* Foetuses with severe malformations that can change the amniotic or urine proteome: complex heart disease, digestive stenosis, fetal immobility.
* Fetus whose mother has chronic infectious diseases (HIV, hepatitis B and C) or acute infectious diseases such chorioamnionitis.
* Parental Refusal.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population will be selected from 31 Multidisciplinary Prenatal Diagnosis Centers
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Renal function (according to Schwartz formula) | month 24
  Renal function (according to Schwartz formula)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane. DECRAMER, MD; PHD, Principal Investigator — Néphrologie pédiatrique - Hôpital des enfants
Locations (31):
- France (31):
  - Hopital Nord, Amiens
  - Chu D Angers, Angers
  - Hopital Saint Jacques, Besançon
  - Hopital Pellegrin, Bordeaux
  - Hopital Morvan, Brest
  - Hopital Femme-Mere-Enfant, Bron
  - Ch Rene Dubos Pontoise, Cergy-Pontoise
  - Hopital Antoine Beclere (Ap Hp), Clamart
  - Chu Estaing, Clermont-Ferrand
  - Hopital Du Bocage, Dijon
  - Chu Grenoble, Grenoble
  - Hopital Jeanne de Flandre, Lille
  - Chu Dupuytren, Limoges
  - Hopital de La Timone (Ap Hm), Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital D'Enfants de Brabois, Nancy
  - Chu de Nantes, Nantes
  - Hopital Lenval, Nice
  - Centre Hospitalier CAREMEAU, Nîmes
  - Hopital Robert Debre, Paris
  - Hopital Armand Trousseau (Ap-Hp), Paris
  - Hopital Necker Enfants Malades (Ap Hp), Paris
  - CHRU De POITIERS LA MILETRIE, Poitiers
  - Hopital Maison Blanche, Reims
  - Hopital Sud, Rennes
  - Hopital Charles Nicole, Rouen
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital de Hautepierre, Strasbourg
  - Maison de Sante Protestante de Bagatelle/Bordeaux, Talence
  - Chu Purpan, Toulouse
  - Hopital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Klein J, Buffin-Meyer B, Boizard F, Moussaoui N, Lescat O, Breuil B, Fedou C, Feuillet G, Casemayou A, Neau E, Hindryckx A, Decatte L, Levtchenko E, Raaijmakers A, Vayssiere C, Goua V, Lucas C, Perrotin F, Cloarec S, Benachi A, Manca-Pellissier MC, Delmas HL, Bessenay L, Le Vaillant C, Allain-Launay E, Gondry J, Boudailliez B, Simon E, Prieur F, Lavocat MP, Saliou AH, De Parscau L, Bidat L, Noel C, Floch C, Bourdat-Michel G, Favre R, Weingertner AS, Oury JF, Baudouin V, Bory JP, Pietrement C, Fiorenza M, Massardier J, Kessler S, Lounis N, Auriol FC, Marcorelles P, Collardeau-Frachon S, Zurbig P, Mischak H, Magalhaes P, Batut J, Blader P, Saulnier Blache JS, Bascands JL, Schaefer F, Decramer S, Schanstra JP; BIOMAN consortium. Amniotic fluid peptides predict postnatal kidney survival in developmental kidney disease. Kidney Int. 2021 Mar;99(3):737-749. doi: 10.1016/j.kint.2020.06.043. Epub 2020 Aug 1. PMID 32750455